CLINICAL TRIAL: NCT03629704
Title: Relationship Between Blood Glucose Variability and Prognosis in Critically Ill Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: KY20170904-06
Record Dates: First submitted 2018-06-18; First posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-06

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Continuous Glucose Monitoring System — Continuous Glucose Monitoring System for 72 hours

SUMMARY:
This study is to evaluate the glycemic variation using Continuous Glucose Monitoring System in patients in the intensive care unit, find out the occult hypoglycemia, and investigate the relationship between glycemic variation, especially the incidence of hypoglycemia and prognosis of patients. Meanwhile, the inflammatory factors were measured and the relationship between inflammatory factors and glycemic variation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with history of diabetes;
2. Patients without history of diabetes, but their random blood glucose≧7.8mmol/L or fast blood glucose≧5 mmol/L;
3. The patients hospitalized in care unit (ICU or CCU) for more than 48 hours.

Exclusion Criteria:

1. Patient had history of mental illness;
2. Patient was not suitable for using the CGMS;
3. blood glucose > 22.2 mmol/L at admission.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted into care unit of Nanjing First Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-08-03 (Estimated); Primary Completion 2018-12-29 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
28 day prognosis | 0-28 days
  Case-fatality at 28 days

SECONDARY OUTCOMES:
Acute Physiology and Chronic Health Evaluation II score | 0-28 days
  Acute Physiology and Chronic Health Evaluation II score
Global registry of acute coronary events risk score | 0-28 days
  Global registry of acute coronary events risk score
Twenty-four-hour mean blood glucose | 1-4 days
  Twenty-four-hour mean blood glucose assessed by CGM
Mean amplitude of glycemic excursion every 24 h | 1-4 days
  Mean amplitude of glycemic excursion every 24 h assessed by CGM
Incidence of hypoglycemia | 1-4 days
  Incidence of hypoglycemia

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Ma, MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University